CLINICAL TRIAL: NCT00268450
Title: A Phase II Study of Neo-Adjuvant Cisplatin, Gemcitabine & Bevacizumab, Followed by Radical Cystectomy for Patients With Muscle Invasive, Resectable, Non-Metastatic Transitional Cell Carcinoma (TCC) of the Bladder
Brief Title: Cisplatin, Bevacizumab, and Gemcitabine Followed by Surgery, Bevacizumab, and Paclitaxel in Treating Patients With Locally Advanced Nonmetastatic Bladder Cancer That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454937; MUSC-AVF-3312; MUSC-HR-15537; GENENTECH-AVF-3312; MUSC-CTO-100892
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-05

CONDITIONS: Bladder Cancer
Keywords: transitional cell carcinoma of the bladder; stage III bladder cancer; stage II bladder cancer; recurrent bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Bevacizumab; Cisplatin; Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- study intervention (Experimental): Neo-adjuvant cisplatin, gemcitabine and bevacizumab followed by radical cystectomy. Patients without residual disease will enter follow up after surgery. Patients with residual disease will receive adjuvant therapy with bevacizumab and ciaplatin.
  Interventions: Biological: bevacizumab; Drug: cisplatin; Drug: gemcitabine hydrochloride; Drug: paclitaxel; Procedure: cysectomy

INTERVENTIONS:
Biological: bevacizumab — Before surgery: given as a 15mg/kg IV over 90 minutes every 21 days for 4 cycles
  After surgery: given as a 15mg/kg IV over 90 minutes every 21 days for 3 cycles
  Other Names: avastin
Drug: cisplatin — Before surgery: given as a 70mg/m2 IV over 60 minutes every 21 days for 4 cycles
Drug: gemcitabine hydrochloride — Before surgery: given as a 1000mg/m2 IV over 30 minutes on days 1 and 8 of a 21 day cycle for 4 cycles
Drug: paclitaxel — After surgery: given as a 175 mg/m2 dose ver 3 hours every 21 days for 3 cycles
Procedure: cysectomy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, gemcitabine, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving combination chemotherapy together with bevacizumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving cisplatin, bevacizumab, and gemcitabine followed by surgery, bevacizumab, and paclitaxel works in treating patients with locally advanced nonmetastatic bladder cancer that can be removed by surgery.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell cancer (TCC) of the bladder

  * Staged as follows:

    * Muscle invasive (T2-T4a)
    * Node negative (N0)

      * No histologically or cytologically proven lymph node metastases
    * Nonmetastatic (M0)

      * No evidence of distant metastases
* Resectable disease
* Able to begin protocol treatment within 6 weeks after transurethral resection and cystoscopic evaluation
* No central nervous system or brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status of 0-2
* Karnofsky 60-100%
* White blood cell count ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* AST(SGOT) and ALT(SGPT) ≤ 2 times upper limit of normal
* Bilirubin ≤1.5 mg/dL
* Creatinine clearance ≥ 60 mL/min
* Urine protein/creatinine ratio < 1.0
* Blood pressure ≤150/100 mm Hg
* No prohibitive medical risks for chemotherapy
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin, gemcitabine hydrochloride, or paclitaxel
* No unstable angina
* No history of myocardial infarction within the past 6 months
* No cardiac arrhythmias
* No New York Heart Association (NYHA) congestive heart failure ≥ grade 2
* No history of stroke within the past 6 months
* No clinically significant peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious nonhealing wound, ulcer, or bone fracture
* No psychiatric illness or other psychosocial situation that would limit ability to comply with study and/or follow-up procedures
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must agree to use adequate contraception prior to study entry and for the duration of study participation
* No significant traumatic injury with in the past 28 days

PRIOR CONCURRENT THERAPY:

* No prior systemic chemotherapy
* No prior pelvic radiation therapy
* More than 4 weeks since prior participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* No concurrent participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* No major surgical procedure or open biopsy within the past 28 days
* No anticipation of need for major surgical procedure during the course of the study
* No minor surgical procedures, fine-needle aspirations, or core biopsies within the past 7 days
* No concurrent treatment with hormones or other chemotherapeutic agents except the following:

  * Steroids given for adrenal failure
  * Hormones administered for nondisease-related conditions (e.g., insulin for diabetes)
  * Intermittent use of dexamethasone as an antiemetic in solid tumor protocols
* No other concurrent investigational or commercial agents or therapies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-09-21 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S. Kraft, MD, Study Chair — Medical University of South Carolina; Gustavo Leone, Study Chair — Medical University of South Carolina, Hollings Cancer Center
Locations (4):
- United States (4):
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Lowcountry Hematology and Oncology, PA, Mt. Pleasant, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Intervention: Neo-adjuvant cisplatin, gemcitabine and bevacizumab followed by radical cystectomy. Patients without residual disease will enter follow up after surgery. Patients with residual disease will receive adjuvant therapy with bevacizumab and ciaplatin.
  bevacizumab: Before surgery: given as a 15mg/kg IV over 90 minutes every 21 days for 4 cycles
  After surgery: given as a 15mg/kg IV over 90 minutes every 21 days for 3 cycles
  cisplatin: Before surgery: given as a 70mg/m2 IV over 60 minutes every 21 days for 4 cycles
  gemcitabine hydrochloride: Before surgery: given as a 1000mg/m2 IV over 30 minutes on days 1 and 8 of a 21 day cycle for 4 cycles
  paclitaxel: After surgery: given as a 175 mg/m2 dose ver 3 hours every 21 days for 3 cycles
  cysectomy
Period: Overall Study
Arm/Group | Study Intervention
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Intervention
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate
Time Frame: From day of first treatment until after cycle 3
Population: Data for this outcome measure was not collected
Arm/Group | Study Intervention
Number analyzed (Participants) | 0

2. Secondary Outcome: Urinary Survivin Levels
Time Frame: Baseline, week 6 and week 12
Population: Data for this outcome measure was not collected
Arm/Group | Study Intervention
Number analyzed (Participants) | 0

3. Secondary Outcome: Urinary Cytogenitics
Time Frame: baseline and week 12
Population: Data for this outcome measure was not collected
Arm/Group | Study Intervention
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival
Time Frame: from first treatment until time of progression or death, whichever comes first
Population: Data for this outcome measure was not collected
Arm/Group | Study Intervention
Number analyzed (Participants) | 0

5. Secondary Outcome: Median Overall Surivial
Time Frame: from first treatment until death
Population: Data for this outcome measure was not collected
Arm/Group | Study Intervention
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Planned Dose Received
Time Frame: from first treatment until end of week 12
Population: Data for this outcome measure was not collected
Arm/Group | Study Intervention
Number analyzed (Participants) | 0

7. Secondary Outcome: Rate of Post-operative Complications
Time Frame: from first treatment until up to 48 hours after surgery.
Population: Data for this outcome measure was not collected
Arm/Group | Study Intervention
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Data not collected for this outcome measure
Arm/Group | Study Intervention
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes